CLINICAL TRIAL: NCT05618158
Title: #4Corners4Health: A Social Media Cancer Prevention Program for Rural Emerging Adults
Brief Title: Cancer Prevention for Young Rural Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); University of Arizona (Other); University of Utah (Other); Colorado State University (Other); University of Colorado, Denver (Other); University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0341/0353; 1R01CA268037-01A1 (NIH); 4R01CA268037-04 (NIH); 5R01CA268037-03 (NIH); 5R01CA268037-02 (NIH)
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: social media; cancer prevention; nicotine use; physical activity; nutrition; sun protection; alcohol use; HPV vaccine; media literacy
MeSH Terms: conditions — Neoplasms; Motor Activity; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Randomized stepped-wedge with four cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 Corners Rural Cancer Prevention (Experimental): Four separate Facebook groups, which provide information via posts within the private groups about cancer risk factors (e.g. reducing alcohol consumption, tobacco use cessation, increasing physical activity), behavioral skills to reduce them, benefits of, social support for, and ways to reduce social/financial costs of cancer prevention, and advice from health care providers to decrease barriers. Posts will seek to improve self- and response-efficacy and perceived risk, and link cancer prevention to personal goals.
  Interventions: Behavioral: 4 Corners Rural Health Cancer Prevention

INTERVENTIONS:
Behavioral: 4 Corners Rural Health Cancer Prevention — Participants, aged 18-26, will join a private Facebook group to participate in the intervention. The group is not viewable to the public, including other Facebook users. Content that focuses on cancer prevention behaviors will be posted twice per day for up to 12 months. Each group will be hosted by a moderator who is responsible for managing the intervention goals and participants' engagement.

SUMMARY:
Young adults aged 18-26 engage in a number of behaviors that increase their risk of developing cancer later in life including sedentary lifestyles, unhealthy eating, nicotine produce us, heavy drinking of alcohol, increased UV exposure, and incomplete uptake of HPV vaccination. A multi-risk factor campaign will be developed to reduce these cancer risk behaviors and delivered to young adults over social media, a popular channel that can reach nearly all young adults. The campaign will be evaluated for effectiveness in a rigorous randomized trial with measures of moderate to vigorous physical activity, healthy eating patterns, nicotine product use, alcohol intake, sunburn prevalence, and HPV vaccination uptake.

DETAILED DESCRIPTION:
Several risk factors are prevalent during early adulthood that can lead to cancer later in life. Emerging adults (EAs) aged 18-26 residing in rural areas of the United States engage in many cancer risk behaviors, especially sedentary lifestyles, poor eating patterns, nicotine product use, excess alcohol intake, infrequent sun protection, and inadequate uptake of the HPV vaccine. This application responds to RFA-CA-20-051, "Social and Behavioral Intervention Research to Address Modifiable Risk Factors for Cancer in Rural Populations." The goal is to improve cancer risk behavioral factors among diverse EAs aged 18-26 living in rural counties in the Four Corners states, a unique, underserved region, using a social media campaign designed with community advisors. EAs, including in rural communities, are heavy consumers of online content, especially over social media, and social media provide responsive, engaging, and low-cost platforms for distributing cancer prevention information with high dissemination potential. But, social media also circulate inaccurate, misleading, and harmful information. The specific aims of this research are to: 1) Develop a social media intervention for diverse EAs in rural communities via a community-engaged process that combines expert advice, user-generated content, and online instruction to communicate about behavioral cancer risks, cancer misinformation, counter marketing, digital and media literacy, and family communication; 2) evaluate the effect of a theory-based social media intervention on moderate to vigorous physical activity (MVPA), healthy eating patterns, nicotine product use, alcohol intake, sunburn prevalence, and HPV vaccination with the diverse population of EAs aged 18-26 in rural counties in AZ, CO, NM, and UT (Four Corners states) recruited from Qualtrics' survey panel and enrolled in a pragmatic randomized trial using a stepped-wedge design in which individual EAs will be randomized to 1 of 4 cohorts and receive the social media feed for varying durations in separate Facebook private groups; 3) test if improvements in EAs' cancer risk knowledge and beliefs, digital and media literacy skills, accurate cancer prevention information, and family communication mediate impact of the social media campaign; and 4) explore whether the impact of the social media campaign differs according to: a) level of EAs' engagement with campaign, b) cancer risk factors, and c) biological sex of the participants (as required by NIH). The research is innovative because it tests a theory-based, multi-risk factor approach to cancer prevention with diverse EAs in rural counties, an under-studied population, in a very popular new media. Social media may reach EAs more than interventions through other community channels (e.g., clinics, schools, and workplaces) and for lower cost in the geographically-dispersed, underserved rural communities in the Mountain West. The overall impact is extremely high because it will aid rural EAs in making informed decisions that reduce cancer risk factors and prevent cancer later in life and help EAs critically evaluate and resist misinformation and marketing that promote cancer risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-26 years old
* Resides in a county coded as RUCC 4-9 in Arizona, Colorado, New Mexico, or Utah
* Able to speak and read English
* Has regular social media engagement
* Accepts screening call from study staff
* Consents to participate

Exclusion Criteria:

* Participated in community engagement activities
* Cannot speak and read English
* Has low or no social media engagement
* Does not accept a screening call from study staff
* Does not consent to participate
* Does not give permission for engagement data to be extracted from Facebook private group
* If biologically female, currently pregnant

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1796 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Baseline
  Participants will self-report minutes per week of moderate to vigorous physical activity.
Physical Activity | 3 months
  Participants will self-report minutes per week of moderate to vigorous physical activity.
Physical Activity | 12 months
  Participants will self-report minutes per week of moderate to vigorous physical activity.
Physical Activity | 24 months
  Participants will self-report minutes per week of moderate to vigorous physical activity.
Diet | Baseline
  Participants will self-report intake per day of fruits, vegetables, whole grains/fiber, added sugars (from sugar-sweetened beverages), and red/processed meats.
Diet | 3 months
  Participants will self-report intake per day of fruits, vegetables, whole grains/fiber, added sugars (from sugar-sweetened beverages), and red/processed meats.
Diet | 12 months
  Participants will self-report intake per day of fruits, vegetables, whole grains/fiber, added sugars (from sugar-sweetened beverages), and red/processed meats.
Diet | 24 months
  Participants will self-report intake per day of fruits, vegetables, whole grains/fiber, added sugars (from sugar-sweetened beverages), and red/processed meats.
Nicotine Product Use | Baseline
  Participants will self-report tobacco/nicotine use in the past 30 days (every day, some days, not at all).
Nicotine Product Use | 3 months
  Participants will self-report tobacco/nicotine use in the past 30 days (every day, some days, not at all).
Nicotine Product Use | 12 months
  Participants will self-report tobacco/nicotine use in the past 30 days (every day, some days, not at all).
Nicotine Product Use | 24 months
  Participants will self-report tobacco/nicotine use in the past 30 days (every day, some days, not at all).
Alcohol Intake | Baseline
  Participants self-report consumption of number of alcoholic drinks in the past 30 days.
Alcohol Intake | 3 months
  Participants self-report consumption of number of alcoholic drinks in the past 30 days.
Alcohol Intake | 12 months
  Participants self-report consumption of number of alcoholic drinks in the past 30 days.
Alcohol Intake | 24 months
  Participants self-report consumption of number of alcoholic drinks in the past 30 days.
Uv Exposure | Baseline
  Participants will self-report number of sunburns.
Uv Exposure | 3 months
  Participants will self-report number of sunburns.
Uv Exposure | 12 months
  Participants will self-report number of sunburns.
Uv Exposure | 24 months
  Participants will self-report number of sunburns.
HPV Vaccination | Baseline
  Participants will self-report whether or not they have received one or more doses of the HPV vaccine.
HPV Vaccination | 3 months
  Participants will self-report whether or not they have received one or more doses of the HPV vaccine.
HPV Vaccination | 12 months
  Participants will self-report whether or not they have received one or more doses of the HPV vaccine.
HPV Vaccination | 24 months
  Participants will self-report whether or not they have received one or more doses of the HPV vaccine.

SECONDARY OUTCOMES:
Physical Activity | Baseline
  Participants will self-report number of minutes per week engaging in physical activity to determine if they meet the 150 minutes per week recommendation.
Physical Activity | 3 months
  Participants will self-report number of minutes per week engaging in physical activity to determine if they meet the 150 minutes per week recommendation.
Physical Activity | 12 months
  Participants will self-report number of minutes per week engaging in physical activity to determine if they meet the 150 minutes per week recommendation.
Physical Activity | 24 months
  Participants will self-report number of minutes per week engaging in physical activity to determine if they meet the 150 minutes per week recommendation.
Diet | Baseline
  Participants will self-report frequency of eating meals away from home/fast food.
Diet | 3 months
  Participants will self-report frequency of eating meals away from home/fast food.
Diet | 12 months
  Participants will self-report frequency of eating meals away from home/fast food.
Diet | 24 months
  Participants will self-report frequency of eating meals away from home/fast food.
Nicotine Product Use | Baseline
  Participants will self-report tobacco/nicotine use in the past 7 days (every day, some days, not at all).
Nicotine Product Use | 3 months
  Participants will self-report tobacco/nicotine use in the past 7 days (every day, some days, not at all).
Nicotine Product Use | 12 months
  Participants will self-report tobacco/nicotine use in the past 7 days (every day, some days, not at all).
Nicotine Product Use | 24 months
  Participants will self-report tobacco/nicotine use in the past 7 days (every day, some days, not at all).
Nicotine Product Use | Baseline
  Participants will self-report readiness to quit using a 10 point rating scale (1=no thought of quitting; 10=taking action to quit).
Nicotine Product Use | 3 months
  Participants will self-report readiness to quit using a 10 point rating scale (1=no thought of quitting; 10=taking action to quit).
Nicotine Product Use | 12 months
  Participants will self-report readiness to quit using a 10 point rating scale (1=no thought of quitting; 10=taking action to quit).
Nicotine Product Use | 24 months
  Participants will self-report readiness to quit using a 10 point rating scale (1=no thought of quitting; 10=taking action to quit).
Alcohol Intake | Baseline
  Participants will self-report number of times binge drinking in the past 30 days.
Alcohol Intake | 3 months
  Participants will self-report number of times binge drinking in the past 30 days.
Alcohol Intake | 12 months
  Participants will self-report number of times binge drinking in the past 30 days.
Alcohol Intake | 24 months
  Participants will self-report number of times binge drinking in the past 30 days.
UV Exposure | Baseline
  Participants will self-report sun protection behaviors with percent of sun exposure hours using sun protection.
UV Exposure | 3 months
  Participants will self-report sun protection behaviors with percent of sun exposure hours using sun protection.
UV Exposure | 12 months
  Participants will self-report sun protection behaviors with percent of sun exposure hours using sun protection.
UV Exposure | 24 months
  Participants will self-report sun protection behaviors with percent of sun exposure hours using sun protection.
HPV Vaccination | Baseline
  Participants will self-report if they have completed the series of HPV vaccination by receiving 3 doses of the vaccine.
HPV Vaccination | 3 months
  Participants will self-report if they have completed the series of HPV vaccination by receiving 3 doses of the vaccine.
HPV Vaccination | 12 months
  Participants will self-report if they have completed the series of HPV vaccination by receiving 3 doses of the vaccine.
HPV Vaccination | 24 months
  Participants will self-report if they have completed the series of HPV vaccination by receiving 3 doses of the vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (5):
- United States (5):
  - University of Arizona, Tucson, Arizona
  - University of Colorado Denver, Aurora, Colorado
  - Colorado State University, Fort Collins, Colorado
  - University of New Mexico, Albuquerque, New Mexico
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Warner EL, Kinsey A, Walkosz BJ, Berteletti J, Nuss K, Small A, Woodall WG, Kepka D, Taren D, Skiba MB, Guest DD, Blair CK, Gordon JS, Wetter DW, Borrayo EA, Henry KL, Sussman AL, Buller DB. A Web-Based Cancer Prevention Intervention for Rural Emerging Adults: Mixed Methods Development and Pilot-Testing Study. J Med Internet Res. 2026 Jan 8;28:e80803. doi: 10.2196/80803. PMID 41505184
- [Derived] Buller DB, Sussman AL, Thomson CA, Kepka D, Taren D, Henry KL, Warner EL, Walkosz BJ, Woodall WG, Nuss K, Blair CK, Guest DD, Borrayo EA, Gordon JS, Hatcher J, Wetter DW, Kinsey A, Jones CF, Yung AK, Christini K, Berteletti J, Torres JA, Barraza Perez EY, Small A. #4Corners4Health Social Media Cancer Prevention Campaign for Emerging Adults: Protocol for a Randomized Stepped-Wedge Trial. JMIR Res Protoc. 2024 Feb 22;13:e50392. doi: 10.2196/50392. PMID 38386396